CLINICAL TRIAL: NCT03082248
Title: Second Opinion in Spinal Surgery Indications: Cost-Effectiveness Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Low Back Pain
Record Dates: First submitted 2017-03-03; First posted 2017-03-17 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2018-07

CONDITIONS: Low Back Pain; Lumbar Spine Injury
Keywords: Low Back Pain; Surgery; Lumbar Spine; Physical Therapy Modalities; Rehabilitation
MeSH Terms: conditions — Low Back Pain; Spinal Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy Group (Other): 10-week supervised physiotherapeutic intervention; all patients will receive educational leaflets and folders for maintenance and adherence to the treatment program.
  Interventions: Other: Physical Therapy
- Spinal Surgery Group (Other): Surgical procedures and techniques specific for the low back region, previously discussed and agreed upon among surgeons according to patients description.
  Interventions: Procedure: Spinal Surgery

INTERVENTIONS:
Other: Physical Therapy — Patients allocated to the conservative treatment group will receive physical therapy according to the treatment-based classification approach and also educational leaflets and folders.
  Arms: Physical Therapy Group
Procedure: Spinal Surgery — Patients allocated to the surgical procedure group will undergo spinal surgery procedures and techniques specific for the low back region.
  Arms: Spinal Surgery Group

SUMMARY:
Low back pain is a common symptom, which often affects the adult population. Studies show that over the past two decades, costs related to spinal surgery have increased significantly, leading to speculation about what would be motivating this phenomenon. Although expenses with physical therapy treatments and less invasive surgical procedures remained relatively stable, the amount spent with more complex spine surgeries increased exponentially until they became the procedures with the highest costs in healthcare. The criteria for surgical indication are not uniform among surgeons and therefore a study of second opinion in spine surgeries is urgently needed. The present study aims to 1) quantify cost-effectiveness of second opinion for patients with spinal surgery indication 2) evaluate effectiveness of conservative and surgical treatment for degenerative diseases of the lumbar spine 3) define objective criteria for indication of conservative and surgical treatment using evidence-based medicine 4) evaluate prognosis of biological markers in the follow-up of patients with lumbar affections 5) evaluate interobserver agreement of physicians in relation to the diagnoses and treatment proposals in patients with diseases of the lumbar spine 6) verify effectiveness of patients who were operated on, compared to patients who were not operated. A prospective cohort study will be conducted, in which patients with an indication of surgical spinal treatment will be evaluated for a second opinion. First evaluation diagnoses and indications for patient treatment will be compared with the second opinion evaluation. All patients who choose to participate on the study will be followed up for a year for evaluations concerning cost-effectiveness, pain, quality of life, function and blood biomarkers. The outcomes will be compared using linear or generalized mixed models and descriptive analyzes of the study population program will be carried out; Statistical agreement will be observed between the first and second opinion and also patient acceptance rates for the treatment proposed in the second indication, evaluating the validity of the project approach. A five-year budget impact analysis will also be carried out, taking into account the population who was eligible for treatment according to the admission flow of a private outpatient setting.

DETAILED DESCRIPTION:
The present study could provide benefits to all aspects of treatment approaches involved in patients with low back pain: for the entire medical community by presenting better information about the actual surgical indications for patients with low back pain; for health insurers and in general, who can spend their investments in really effective areas, and especially for patients, who will receive appropriate treatments for their conditions.

190 patients with indication of surgical treatment will be enrolled for this clinical trial and will be advised to receive a second opinion at Hospital Israelite Albert Einstein (HIAE).

Both assessments (with orthopedic physicians) will be compared, and when consensus is reached about diagnostic hypotheses and treatment, patients will be referred for conservative or surgical treatment. Any disagreements will be resolved by a committee of spine surgeons (four orthopedists and four neurosurgeons with more than 15 years of experience).

When the treatment chosen for the first medical care (two consultations of the orthopedic surgeons) is the conservative treatment, patients will be referred to consultations in the rehabilitation center. When surgical treatment is indicated, the patient will be referred to one of the eight surgeons of the spinal committee.

All patients will have the freedom of choice to decide to participate in the study guided by the second opinion service or perform the recommended treatment in the first hospital in which they were treated.

Sample size: For the calculation of the sample size estimate, we considered data presented in the study by van der Roer et al. (2006), in which the mean score obtained by the EuroQol instrument in pre-treatment patients was 0.70 in chronic patients, with standard deviation of 0.19. Assuming that the correlation between the measurements obtained at the two main moments of comparison (baseline and after 10 weeks of treatment) is of the order of 0.5 and that the minimally relevant difference between the two moments is 0.07, we estimate that 90 patients should be considered in the conservative treatment group. Assuming that of the patients who use the second opinion service about 55% will perform surgical procedures in the service, we estimate that 100 patients should be included in this group. Sample size estimates were performed with the statistical package STATA version 10.0, considering 90% power and 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with surgery indication (referred by the health care provider) for the treatment of degenerative diseases of the lumbar spine (basically: intervertebral disc disease, degenerative spondylolisthesis, lumbar canal stenosis, facet low back pain and lumbar instability);
2. no contraindication to general anesthesia or any physiotherapeutic procedure;
3. able to understand Portuguese language and after acceptance of a written consent.

Exclusion Criteria:

* Patients with:

  1. spinal fractures;
  2. scoliosis greater than 20 degrees;
  3. congenital deformities;
  4. spinal tumors;
  5. confirmed or suspected pregnancy;
  6. history of previous surgery in the spine; and,
  7. unable to participate in the follow-up (due to inability to read or complete the required forms).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Cost Effectiveness analysis | 12 months after treatment
  EuroQoL will be combined with a Visual Analogue Scale(VAS) to carry out the cost-effectiveness analysis of the second opinion program.

SECONDARY OUTCOMES:
Change in Pain Intensity | 1, 3, 6 and 12 months after treatment
  Pain intensity will be measured using VAS 0-10 (0 being no pain and 10 maximum pain)
Change in Disability | 1, 3, 6 and 12 months after treatment
  Disability will be measured by the Oswestry Disability Index, Brazilian version 2.0.
Change in Global Impression of Recovery | 1, 3, 6 and 12 months after treatment
  Global impression of recovery will be measured by the Global Perceived Effect of Change(GPE)
Change in Kinesiophobia | 1, 3, 6 and 12 months after treatment
  Assessment of fear avoidance beliefs related to physical activity and work will be evaluated by the questionnaire Fear avoidance Beliefs Questionnaire (FABQ)
Change in Psychosocial Risk Prognosis | 1, 3, 6 and 12 months after treatment
  Psychosocial risk prognosis will be measured by the brazilian version of the STarT Back screening tool
Change in Mood Disorders in The setting of Medical Practice | 1, 3, 6 and 12 months after treatment
  Anxiety and depression aspects will be measured by the Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ferretti, MD, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We are happy to share our data with researchers that would like to use it on an individual participant data

REFERENCES:
- [Background] Martin BI, Deyo RA, Mirza SK, Turner JA, Comstock BA, Hollingworth W, Sullivan SD. Expenditures and health status among adults with back and neck problems. JAMA. 2008 Feb 13;299(6):656-64. doi: 10.1001/jama.299.6.656. PMID 18270354
- [Background] Dagenais S, Caro J, Haldeman S. A systematic review of low back pain cost of illness studies in the United States and internationally. Spine J. 2008 Jan-Feb;8(1):8-20. doi: 10.1016/j.spinee.2007.10.005. PMID 18164449
- [Background] Healy WL, Peterson RN. Department of Justice investigation of orthopaedic industry. J Bone Joint Surg Am. 2009 Jul;91(7):1791-805. doi: 10.2106/JBJS.I.00096. No abstract available. PMID 19571103
- [Background] Perret D, Rosen C. A physician-driven solution--the Association for Medical Ethics, the Physician Payment Sunshine Act, and ethical challenges in pain medicine. Pain Med. 2011 Sep;12(9):1361-75. doi: 10.1111/j.1526-4637.2011.01217.x. PMID 21914121
- [Background] Viola DC, Lenza M, Almeida SL, Santos OF, Cendoroglo Neto M, Lottenberg CL, Ferretti M. Spine surgery cost reduction at a specialized treatment center. Einstein (Sao Paulo). 2013 Jan-Mar;11(1):102-7. doi: 10.1590/s1679-45082013000100018. PMID 23579752
- [Background] Delitto A, Erhard RE, Bowling RW. A treatment-based classification approach to low back syndrome: identifying and staging patients for conservative treatment. Phys Ther. 1995 Jun;75(6):470-85; discussion 485-9. doi: 10.1093/ptj/75.6.470. PMID 7770494
- [Background] Fritz JM, Cleland JA, Childs JD. Subgrouping patients with low back pain: evolution of a classification approach to physical therapy. J Orthop Sports Phys Ther. 2007 Jun;37(6):290-302. doi: 10.2519/jospt.2007.2498. PMID 17612355
- [Background] van der Roer N, Ostelo RW, Bekkering GE, van Tulder MW, de Vet HC. Minimal clinically important change for pain intensity, functional status, and general health status in patients with nonspecific low back pain. Spine (Phila Pa 1976). 2006 Mar 1;31(5):578-82. doi: 10.1097/01.brs.0000201293.57439.47. PMID 16508555